CLINICAL TRIAL: NCT05377346
Title: A Comparison of the Effect of Paratracheal and Cricoid Pressure on the Placement of the I-gel.
Brief Title: Effect of Paratracheal and Cricoid Pressure on the Placement of the I-gel.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202205
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Paratracheal Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paratracheal pressure group (Experimental): After the induction of anesthesia, the i-gel is placed under the application of paratracheal pressure.
  Interventions: Other: Placement of the i-gel
- Cricoid pressure group (Active Comparator): After the induction of anesthesia, the i-gel is placed under the application of cricoid pressure.
  Interventions: Other: Placement of the i-gel

INTERVENTIONS:
Other: Placement of the i-gel — The lubricated i-gel is inserted into the mouth and introduced along the hard palate with a continuous and gentle push until resistance was felt in the hypopharynx.

SUMMARY:
This study aims to compare the effect of paratracheal and cricoid pressure on placement of the i-gel in terms of the success rate of i-gel insertion, time to placement, the rate of optimal position of the device, and difficulty of i-gel placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Presence of an upper airway anatomic variation or pathology
* Increased risk of pulmonary aspiration
* Known or predicted difficult airway
* Surgery requiring lateral or prone position, head and neck surgery
* Requirements for postoperative ventilator care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
The success rate of the i-gel placement | Immediately after the placement of the i-gel
  Successful placement of the i-gel is determined by proper chest expansion, the presence of a square waveform on the capnogram, absence of an audible leak, and lack of gastric insufflations.

SECONDARY OUTCOMES:
Time to placement of the i-gel | Immediately after the placement of the i-gel
  Time to placement is defined as the time from picking up the i-gel to observing the end-tidal CO2 waveform.
The rate of optimal position of the i-gel | Immediately after the placement of the i-gel
  The anatomic position of the device is evaluated using a fiberoptic bronchoscope and graded on a scale of 1-4 as follows: 4, only the vocal cords seen; 3, vocal cords and posterior part of the epiglottis seen; 2, vocal cords and anterior part of the epiglottis seen; 1, vocal cords not seen, but adequate ventilation
Difficulty of the i-gel placement | Immediately after the placement of the i-gel
  Difficulty of the i-gel placement is assessed as follows; 1, very easy; 2, easy; 3, moderate; 4, difficult; 5. very difficult
Tidal volume | At 1 minute after the placement of the i-gel
  Tidal volume is assessed with or without each pressure using the ventilator setting (volume-control mode with a tidal volume of 8 mL/kg of ideal body weight, respiratory rate of 12 breaths/min, and zero end-expiratory pressure).
Peak inspiratory pressure | At 1 minute after the placement of the i-gel
  Peak inspiratory pressure is assessed with or without each pressure using the ventilator setting (volume-control mode with a tidal volume of 8 mL/kg of ideal body weight, respiratory rate of 12 breaths/min, and zero end-expiratory pressure)..

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Won D, Kim H, Chang JE, Lee JM, Kim TK, Kim H, Min SW, Hwang JY. Comparison of the effects of paratracheal pressure and cricoid pressure on placement of the i-gel(R) supraglottic airway: a randomized clinical trial. Can J Anaesth. 2024 Jul;71(7):996-1003. doi: 10.1007/s12630-024-02741-1. Epub 2024 Mar 20. PMID 38507025